CLINICAL TRIAL: NCT04272463
Title: ChAracterisation of ItaliaN Severe Uncontrolled Asthmatic patieNts Key Features When Receiving Benralizumab in a Real Life Setting: an Observational rEtrospective Study
Brief Title: ChAracterisation of ItaliaN Severe Uncontrolled Asthmatic patieNts Key Features When Receiving Benralizumab
Acronym: ANANKE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00073
Record Dates: First submitted 2020-01-19; First posted 2020-02-17 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: No intervention — Patients currently in treatment with benralizumab as per approved indication and clinical practice

SUMMARY:
This is an observational, Italian multi-center, retrospective cohort study with enrollment visit on patients suffering from severe eosinophilic asthma who started benralizumab in the Sampling Program or as per normal clinical practice in Italy.

DETAILED DESCRIPTION:
A retrospective cohort study design involving secondary data collection was chosen to appropriately address the primary objective in a relatively short period of time after enrollment phase initiation: in fact, since the Italian Sampling Program on benralizumab was active since July 2018, clinical data on patients exposed to benralizumab are already available. No treatments will be administered per protocol requirement, but instead according to normal clinical practice; since benralizumab first administration occurs before inclusion in the study (as per chosen study design), the decision to include the patient in the study is clearly separated from the prescription of benralizumab, in accordance with the observational nature of the study. In order to be eligible for the study, for each patient, the index date shall be at least 3 months prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥18 years) at the start of benralizumab treatment within the sampling program or per clinical practice ("index date").
2. Patients with severe eosinophilic asthma requiring a stable treatment of high doses of inhaled corticosteroids and a long acting β2 agonist ± additional asthma controller (according to clinician's judgment).
3. Patients who started benralizumab and received at least one injection at least 3 months before enrollment, either within the sampling program or as per routine clinical practice.
4. Patients who signed the informed consent and privacy form at enrollment visit.
5. Patients with available hospital medical chart since the start of benralizumab treatment within the sampling program or per clinical practice ("index date").

Exclusion Criteria:

1. Patients who, during the observation period, received benralizumab in a clinical experimental trial.
2. Patients who, during the observation period, participated in studies imposing a specific patient's management strategy which does not correspond to the site's normal clinical practice.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll patients with severe eosinophilic asthma treated with benralizumab. Patients can be enrolled if they received benralizumab either within the sampling program or as per routine clinical practice.
  Participating sites will enroll patients in a consecutive manner when patients come for their regular visit, in order to minimize the risk of selection bias.
  A total of 200 patients are expected to be included in the study by around 20 sites, corresponding to approximately 10 patients/site: it is estimated that the study will enroll approximately 25 patients per month in the around 20 centers involved (approximately 1.3 patients/month/center). This target sample size is expected to be reached durin
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
key features at benralizumab treatment start) | At baseline
  Total IgE and eosinophils count in peripheral blood as measured at index date Lung function assessments Presence of comorbidities Previous severe exacerbations in the 12 months before index date. Previous treatments with biologics for asthma before index date. Maintenance asthma treatment(s) ongoing at index date.

SECONDARY OUTCOMES:
severe exacerbations during benralizumab treatment | at 16 weeks
  Proportion of patients experiencing at least 1 severe exacerbation during benralizumab treatment.
  Severe exacerbation incidence rate during benralizumab treatment, calculated as the number of patients with at least one exacerbation occurred during benralizumab treatment (cases) divided by the person-time at risk considering the duration of observation while the patient was receiving benralizumab.
  Annual severe exacerbation rate, which will be calculated as the ratio between the total number of severe exacerbations occurred in the sample and the total number of person-years (i.e. the actual time-at-risk that all evaluable patients contributed to the study while they were in treatment with benralizumab).
ICS and OCS change during benralizumab treatment | at 16 weeks
  ICS dose change of any extent Change of OCS dose (final dose* with respect to index date; if applicable)
IgE and eosinophils count during benralizumab treatment, and changes over time with respect to benralizumab treatment start | at 16 weeks
  Descriptive statistics of total IgE and eosinophils count in peripheral blood as measured at the time points specified.
  Descriptive statistics of intra-patient changes over time in total IgE and eosinophils count in peripheral blood, at each time points specified with respect to index date (according to data availability).
lung function parameters during benralizumab treatment, and changes over time with respect to benralizumab treatment start | at 16 weeks
  Descriptive statistics of lung function parameters as measured at the time points specified.
  Descriptive statistics of intra-patient changes over time in lung function parameters, at each time points specified with respect to index date (according to data availability).
patients' asthma control level and quality of life at benralizumab treatment start, during the observation period, and changes over time with respect to benralizumab treatment start | at 16 weeks
  Descriptive statistics of Asthma Control Test (ACT) total score at index date (if available).
  Descriptive statistics of ACT total score at the time points specified in chapter 4.2 (according to data availability), along with proportion of patients with well-controlled asthma (i.e. ACT score major of 20).
  Descriptive statistics of intra-patient changes in ACT total score, at each time points specified in chapter 4.2 with respect to index date (according to data availability).
  Descriptive statistics of Asthma Quality of Life Questionnaire (AQLQ) total score at index date (if available).
  Descriptive statistics of AQLQ total score at the time points specified in chapter 4.2 (according to data availability).
  Descriptive statistics of intra-patient changes in AQLQ total score, at each time points specified in chapter 4.2 with respect to index date (according to data availability).
patient's adherence to benralizumab treatment | at 16 weeks
  Descriptive statistics of level of patient's adherence to benralizumab treatment, computed as the ratio (in percentage) between the number of actual injections received during the observation period over the number of expected injections (which will be estimated considering the injection schedulation specified in the SmPC).
healthcare resource utilization during benralizumab treatment | at 16 weeks
  Descriptive statistics of total number (per patient) of the following healthcare resource utilization occurred during benralizumab treatment: GP/specialist visits for asthma, ER admissions for asthma, and hospitalizations for asthma.
benralizumab discontinuation | at 16 weeks
  Proportion of patients with benralizumab permanent discontinuation during the observation period, and description of reasons.
biologic treatments during the observation period | at 16 weeks
  Proportion of patients with subsequent biologic treatments for asthma, and description of type of treatment and reason for switch

CONTACTS AND LOCATIONS:
Overall Officials: Girolamo Pelaia, MD, Principal Investigator — Università degli Studi Magna Graecia; Pietro Bracciale, MD, Principal Investigator — Ospedale di Ostuni; Francesco Menzella, MD, Principal Investigator — Arcispedale Santa Maria Nuova, Reggio Emilia; Giorgio W Canonica, MD, Principal Investigator — Humanitas University Rozzano; Andrea Matucci, MD, Principal Investigator — AO Careggi Firenze; Mariella D'Amato, MD, Principal Investigator — AO Dei Colli Monaldi Napoli; Elisabetta Romagnoli, MD, Principal Investigator — Treviso Regional Hospital; Fausto De Michele, MD, Principal Investigator — AO Cardarelli Napoli; Paolo Palange, MD, Principal Investigator — Policlinico Umberto I Roma; Adriano Vaghi, MD, Principal Investigator — AO Garbagnate Milanese; Pietro Schino, MD, Principal Investigator — Ospedale Miulli, Acquaviva delle Fonti; Paola Rogliani, MD, Principal Investigator — University of Rome Tor Vergata; Elena Bargagli, MD, Principal Investigator — Policlinico Le Scotte Siena; Stefano Centanni, MD, Principal Investigator — Ospedale San Paolo Milano; Cristiano Caruso, MD, Principal Investigator — IRCCS Fondazione Gemelli Roma; Stefano Del Giacco, MD, Principal Investigator — Ospedale Monserrato Cagliari; Maria Aliani, MD, Principal Investigator — IRCCS Maugeri Cassano delle Murge; Diego Bagnasco, MD, Principal Investigator — IRCCS San Martino Genova; Antonino Musarra, MD, Principal Investigator — Casa della Salute Scilla; Fabiano Di Marco, MD, Principal Investigator — Ospedale Papa Giovanni XXIII Bergamo; Gianenrico Senna, MD, Principal Investigator — Ospedale Borgo Trento - Verona; Luigi Macchia, MD, Principal Investigator — Policlinico Bari
Locations (18):
- Italy (18):
  - Research Site, Acquaviva delle Fonti
  - Research Site, Bergamo
  - Research Site, Cassano Murge
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Garbagnate Milanese
  - Research Site, Milan
  - Research Site, Monserrato
  - Research Site, Napoli
  - Research Site, Ostuni
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Siena
  - Research Site, Torino
  - Research Site, Treviso
  - Research Site, Verona

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Canonica GW, Consani L, Malerba L, Pelaia G, Vultaggio A; ANANKE investigators. Effects of benralizumab in patients with severe eosinophilic asthma (SEA): A plain language summary of the ANANKE study. Immunotherapy. 2024;16(14-15):913-923. doi: 10.1080/1750743X.2024.2386899. Epub 2024 Sep 17. PMID 39287158
- [Derived] Vultaggio A, Aliani M, Altieri E, Bracciale P, Brussino L, Caiaffa MF, Cameli P, Canonica GW, Caruso C, Centanni S, D'Amato M, De Michele F, Del Giacco S, Di Marco F, Menzella F, Pelaia G, Rogliani P, Romagnoli M, Schino P, Senna G, Benci M, Boarino S, Schroeder JW. Long-term effectiveness of benralizumab in severe eosinophilic asthma patients treated for 96-weeks: data from the ANANKE study. Respir Res. 2023 May 20;24(1):135. doi: 10.1186/s12931-023-02439-w. PMID 37210543
- [Derived] Menzella F, Bargagli E, Aliani M, Bracciale P, Brussino L, Caiaffa MF, Caruso C, Centanni S, D'Amato M, Del Giacco S, De Michele F, Di Marco F, Pastorello EA, Pelaia G, Rogliani P, Romagnoli M, Schino P, Senna G, Vultaggio A, Simoni L, Ori A, Boarino S, Vitiello G, Altieri E, Canonica GW. ChAracterization of ItaliaN severe uncontrolled Asthmatic patieNts Key features when receiving Benralizumab in a real-life setting: the observational rEtrospective ANANKE study. Respir Res. 2022 Feb 19;23(1):36. doi: 10.1186/s12931-022-01952-8. PMID 35183167
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00073&attachmentIdentifier=9c02d35c-2d0a-4a54-bc58-69278ad0a975&fileName=D3250R00073_CSR_Synopsis.pdf&versionIdentifier=